CLINICAL TRIAL: NCT03003039
Title: A Study Comparing GB241 And Rituximab in Patients With B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Yoko Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GB241NHL1
Record Dates: First submitted 2016-12-20; First posted 2016-12-26 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: B-Cell Lymphoma
Keywords: GB241; Rituximab; B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GB241 (Experimental): GB241:375 mg/m2, iv, one infusion
  Interventions: Biological: GB241
- Rituximab (Active Comparator): Rituximab: 375 mg/m2, iv, one infusion
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: GB241 — Single intravenous infusion (IV) 375 mg/m2
  Arms: GB241
Biological: Rituximab — Single intravenous infusion (IV) 375 mg/m2
  Arms: Rituximab

SUMMARY:
The purpose of this study is the area under the curve (AUC) for GB241 and rituximab concentrations.

ELIGIBILITY:
Inclusion Criteria:

* having histologically confirmed NHL expressing CD20 antigen
* having obtained CR (complete remission) or CRu (uncertain complete remission) after the prior therapy
* signed an informed consent form which was approved by the institutional review board of the respective medical center
* aged from 18 to 75 years
* ECOG performance status of 0 to 1
* expected survival of at least ≥ 3 months

Exclusion Criteria:

* had received rituximab or other anti-CD20(+) monoclonal antibody treatment within 1 year before enrollment
* having to be at least 4 weeks beyond prior anticancer therapy including corticosteroid, or have not recovered from significant toxicities of prior therapy
* participating in other clinical trial within 30 days before enrolment
* with serious hematologic dysfunction (white blood cell count of <3.0×103/uL; absolute neutrophil count of <1.5×103/ uL; platelet count of < 75×103/uL; hemoglobin level of < 8.0 g/dL); hepatic dysfunction (total bilirubin level of > 1.5×ULN; aspartate amino transferase (AST) and alanine amino transferase (ALT) levels of >2.5 × ULN; renal dysfunction (serum creatinine level of > 1.5×ULN ); and International normalized ratio (INR) and partial thromboplastin time or activated partial thromboplastin time (aPTT) > 1.5 × ULN (unless on therapeutic coagulation)
* had received live vaccine within 4 weeks prior to study entry
* with other malignancies ; or central nervous system (CNS) lymphoma, AIDS-related lymphoma; or active opportunistic infection, a serious nonmalignant disease
* seropositive for HCV antibody, or HIV antibody, or hepatitis B virus surface antigen (HBsAg). HBc antibody seropositive, but HBV DNA and HBsAg negative patients may participle following consultation with a hepatitis expert regarding monitoring and use of HBV antiviral therapy, and provided they agree to receive treatment as indicated
* recent major surgery (within 28 days prior to study entry )
* with a history of allergic reaction or protein product allergy including murine proteins
* pregnant or lactating or not accepted birth control methods including male patients
* patients considered unsuitable by PI
* previous malignant tumor except cured cervical cancer,basal cell carcinoma and squamous cell skin cancer
* active opportunistic infections and other serious non neoplastic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) for GB241 and rituximab concentrations | 85 days

SECONDARY OUTCOMES:
AUC for GB241 and rituximab concentrations | 1 week, 2 weeks, 4 weeks, 8 weeks and 12 weeks
Maximum observed concentration of the GB241 and rituximab | 85 days
Degree of clearance from baseline of CD19+ , CD20+ B-cells between the two study arms | 85 days
Comparison of AEs between the two study arms | 85 days
Comparison of the incidence rate of HACA（host anti-chimeric antibody） between the two study arms | 85 days

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China